CLINICAL TRIAL: NCT01744977
Title: Evaluate the Efficacy, Perceptions and Cost of an Innovative Cholesterol Packaging
Brief Title: Cholesterol Medication Packaging Study
Acronym: MWV_CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 01642
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Product Packaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adherence Packaging Intervention Group (Experimental): [MeadWestvaco Packaging Intervention Arm] At baseline, the intervention arm will receive instructions from the RA on obtaining medication refills and the first fill of their statin medication from the VA pharmacy. At this time, the pharmacist will provide counseling including 1) use of adherence packaging, 2) to only use statin medications from the adherence packaging 3) purpose of LDL-related medications 4) how to take the medications.
  Interventions: Behavioral: packaging
- Education Only Group (No Intervention): Control Arm patients will receive primary care and LDL management according to the discretion of their provider. At baseline, patients will receive similar written information on how to obtain medication refills and the importance of taking their cholesterol medications as prescribed. The 6-month interval was selected to maintain contact with patients.

INTERVENTIONS:
Behavioral: packaging — Intervention provides usual statin medication dispensed in pre-prepared adherence packaging (blister packaging) rather than the previously received prescription bottles
  Arms: Adherence Packaging Intervention Group

SUMMARY:
The purpose of the overall study is to improve medication use rates among veterans by looking at the risk factors of low-density lipoprotein cholesterol (LDL). It will involve patients who have high LDL-C level (<130mg/dl) and /or may have difficulty taking their medications based on how often they refilled their medications in the last 12 months.

The investigators will test an innovative adherence packaging relative to usual care. The primary hypothesis is that veterans who receive the intervention will have greater improvement in their medication adherence as measured by pill refill at 6 and 12 months of follow up as compared to the control group.

DETAILED DESCRIPTION:
A sample of participants with elevated LDL level >130 mg/dl and/or <80% medication position ratio in the last 12 months (n=250) will be consented. The study sample will consist of both male and female subjects. Research assistants (RA's) will complete a baseline assessment and then randomly allocated participants to one of the following two groups:

* MeadWestvaco (MWV) Packaging Intervention. Patients randomized to the intervention group will receive the MWV medication adherence packaging and adherence education (Packaging Education.) at baseline from a research pharmacist. The participant will then receive their prescribed cholesterol medication in the MWV packaging over the next 12 months.
* The Education only Group - Patients randomized to the control group will receive educational material about LDL reduction at baseline.

The study includes the following contacts with participants.

* Recruitment letter
* Telephone screening
* Baseline consent and interview - In person for all participants [Only Adherence Packaging Intervention participants will receive baseline discussion and education from the research pharmacist]
* 6 month outcome assessment follow-up - In person for all participants
* 12 month outcome assessment follow-up - In person for all participants
* 12 month phone interview - Optional recorded qualitative interview for intervention participants only.

All participants enrolled in study will be followed for 12 months.

The study includes the following contacts with providers

• Baseline consent and explanation of the adherence packaging - In person for all providers (group style visit)

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in one of three Durham VA Medical Center (DVAMC) Primary Care clinics for at least one year
* AT least one visit to a primary care provider at the Raleigh Community Based Outpatient Clinic (CBOC) or DVAMC associated primary care clinics in the previous 12 months
* Outpatient diagnostic code for hypercholesterolemia
* uncontrolled LDL in the last 12 months and/or poor LDL refill defined as <80% medication adherence in the last 12 months
* prescribed whole tablets of simvastatin, rosuvastatin or pravastatin

Exclusion Criteria:

* Diagnosis of metastatic cancer.
* Active diagnosis of dementia documented in medical record.
* Active diagnosis of psychosis documented in medical record with admission with last 30days.
* Treated with dialysis
* Hospitalized for a stroke, myocardial infarction, coronary artery revascularization in past month.
* Severely impaired hearing, speech or sight. (Patients must be able to respond to phone calls and review adherence literature)
* Participating in another on-going cardio- vascular disease (CVD) risk management study (i.e., pharmaceutical trial or behavioral intervention)
* Does not have access to a telephone
* Resident in nursing facility that manages patients medications or
* Receiving home health care for extended period (home health service for limited time period will not exclude, i.e. scheduled surgical procedure not expected to require care for longer than 30 days)
* Planning to leave the area prior to the anticipated end of participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-12; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hayden B Bosworth, PhD, Principal Investigator — Duke University Medical Center/Durham VA Medical Center, Health Services and Development
Locations (2):
- United States (2):
  - Durham VAMC, Durham, North Carolina
  - Raleigh Community-based Outpatient Clinic (CBOC- Raleigh), Raleigh, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Adherence Packaging Intervention Group: [MeadWestvaco Packaging Intervention Arm] At baseline, the intervention arm will receive instructions from the RA (Research Assistant) on obtaining medication refills and the first fill of their statin medication from the VA pharmacy. At this time, the pharmacist will provide counseling including 1) use of adherence packaging, 2) to only use statin medications from the adherence packaging 3) purpose of LDL-related medications 4) how to take the medications.
  packaging: Intervention provides usual statin medication dispensed in pre-prepared adherence packaging (blister packaging) rather than the previously received prescription bottles
- Education Only Group: Control Arm patients will receive primary care and LDL management according to the discretion of their provider. At baseline, patients will receive similar written information on how to obtain medication refills and the importance of taking their cholesterol medications as prescribed.
Period: Overall Study
Arm/Group | Adherence Packaging Intervention Group | Education Only Group
Started | 120 | 120
6 Month Completed | 113 | 115
Completed | 109 | 115
Not Completed | 11 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — No longer meets inclusion | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adherence Packaging Intervention Group | Education Only Group | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.9) | 62.9 (8.6) | 62.6 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 109 | 110 | 219
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 47 | 41 | 88
  African American or Other | 73 | 79 | 152
Region of Enrollment [Number; unit: participants]
  United States | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: Cholesterol Medication Adherence
Description: Pill refill obtained at 12 months to review change in cholesterol medication adherence over the 12 month period between groups
Time Frame: 12 months
Population: Data on pill refill could not be obtained for 2 of the education only participants.
Measure: Median (Inter-Quartile Range); unit: adherence proportion
Arm/Group | Adherence Packaging Intervention Group | Education Only Group
Number analyzed (Participants) | 120 | 118
adherence proportion | .99 [0.74 to 0.99] | .94 [0.60 to 1.00]
Statistical Analysis 1: Comparison: Adherence Packaging Intervention Group vs Education Only Group; Test type: Non-Inferiority or Equivalence — With an assumed adherence proportion in the Control arm of 0.50, there is 80% power to detect a difference between Control and the intervention arms of 17% or more with 125 patients in each arm; p = 0.300, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in LDL Cholesterol Level as Measured at Baseline, 6months, 12months
Description: obtain non-fasting lipid panel at timepoints to review change in LDL cholesterol levels over the 12 month period (at baseline, 6 and 12 months)
Time Frame: Baseline, 6months, 12months
Population: Cholesterol values could not be obtained for all patients at all time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adherence Packaging Intervention Group | Education Only Group
Number analyzed (Participants) | 120 | 120
mg/dL
  Baseline (n=120/119) | 110.1 (38.8) | 111.6 (31.7)
  6 months (n=112/115) | 101.1 (29.4) | 105.8 (32.8)
  12 months (n=109/115) | 101.3 (34.3) | 102.9 (33.1)
Statistical Analysis 1: Comparison: Adherence Packaging Intervention Group vs Education Only Group; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.839, Mixed Models Analysis — As measured at 12m; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-8.0 to 6.5] — This value summarizes the full 12 month period so Mean Difference (Final Values) is appropriate

ADVERSE EVENTS:
Time Frame: During 1 year study participation
Description: Patients were asked about adverse events at each follow-up appointment and a systematic review of the medical record was completed at each follow-up as well.
Arm/Group | Adherence Packaging Intervention Group | Education Only Group
Serious Adverse Events (participants affected / at risk) | 33/120 | 26/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adherence Packaging Intervention Group (N=120) | Education Only Group (N=120)
Bee Sting- Emergency Room Visit (General disorders) | 0 (0) | 1 (1) — Bee sting
Bleeding- Emergency Room Visit (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Heavy bleeding accompanied by lightheadedness
Cardiac Related Hospitalization or Visit (Cardiac disorders) | 9 (13) | 5 (6) — Includes: chest pain, MI, heart failure, hospitalization including surgery
Bowel Obstruction- Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalization
General Hospitalization (General disorders) | 0 (0) | 1 (1) — chemotherapy complication
Hospitalization-Infection (Infections and infestations) | 1 (1) | 0 (0) — Sepsis related to kidney failure
Hospitalization-Renal (Renal and urinary disorders) | 0 (0) | 1 (1) — Increased Cr, acute renal failure
Hospitalization- Respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Includes: pneumonia, lung disease
Hospitalization-Stroke (Vascular disorders) | 1 (1) | 0 (0)
Musculoskeletal Surgery (Surgical and medical procedures) | 2 (2) | 0 (0) — Knee Arthroplasty Surgery
Death unrelated to study protocol (General disorders) | 2 (2) | 3 (3) — Unrelated pt deaths (cancer, CHF complications, not specified)
Hospitalization-Gastrointestinal (Gastrointestinal disorders) | 1 (1) | 1 (1) — Events include: small bowel obstruction and diverticulitis
Hospitalization-General (General disorders) | 2 (2) | 3 (5) — Events include: Re-occurring treatment for prior dx (spinal injury), Multi-factorial hospitalization causes, MVA events, & Unspecified causes
Hospitalization-Infection (Infections and infestations) | 3 (3) | 3 (4) — Events include: Fever during radiation treatment, Febrile Neutropenia, Cellulitis, Fainting, Food poisoning, UTI
Hospitalization-Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) — Events include: Assault, Spinal surgery rehab, Fractures,
Hospitalization-Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Events include: Lymphadenopathy sarcoma
Hospitaliztion- Nervous (Nervous system disorders) | 0 (0) | 1 (1) — Events include: spinal cord injury biopsy
Hospitalizations-Psychiatric (Psychiatric disorders) | 3 (4) | 1 (1) — Events include: Psychiatric events (due to HIPAA can not collect/provide details)
Hospitalization- Renal (Renal and urinary disorders) | 3 (3) | 1 (1) — Events include: Renal failure, hematuria, Acute kidney disease
Hospitaliztion- Respiratory (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 0 (0) — Events include: Pneumonia, Lung Mass, Impaired gas exchange, pulmonary embolism
Surgery during Hospitaliztion (Surgical and medical procedures) | 11 (12) | 9 (11) — Event include:renal biopsy, amputation (and revision), coronary angiograph, lesion, lung removal, spinal cord bx, spinal surgery, carotid endarterectomy, tendon repair, tumor, nephrectomy, back surgery, hip arthroplasty, cath, appendix, etc
Hospitalization- Vascular (Vascular disorders) | 2 (2) | 1 (1) — Events include: Stroke, Blood clot
Renal blockage- ER Visit (Renal and urinary disorders) | 1 (1) | 0 (0) — Events include: Blocked catheter,
Bronchitis/COPD- ER Visit (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pt came to ER for SOB via EMS.
Scheduled Outpatient Surgery (General disorders) | 2 (2) | 1 (1) — Events include: laryngoscopy with lesion removal, thyroid nodule
Scheduled Outpatient Surgery- Renal (Renal and urinary disorders) | 1 (2) | 0 (0) — Events include: PCN placement for ureteral obstruction, bladder tumor resection,
Planned outpatient surgery- Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Rotator cuff repair

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No